CLINICAL TRIAL: NCT01587092
Title: WorkStation Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBRC 12015
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Sedentary Lifestyle
Keywords: walking; physical activity; sedentary behavior; workplace
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Working Condition Group (Placebo Comparator): Participants assigned to the usual working condition control group will continue to work in their usual environment and accustomed manner. The control group participants will have access to the Workstations at the completion of study.
  Interventions: Behavioral: Usual Working Condition
- WorkStation Intervention Group (Active Comparator): Participants will be asked to walk for up to 1.5 hours per day on the treadmill. This will be split into two 45 minute sessions per day. Behavioral support will focus on adherence to frequency (attending scheduled sessions). Participants self-select speed of walking and time (they have up to 45 minutes allotted, but may choose less as they like).
  Interventions: Behavioral: WorkStation

INTERVENTIONS:
Behavioral: WorkStation — Participants will be asked to attend 2 scheduled sessions per day of treadmill walking, which will replace their sitting desk time. Participants will complete 2 sessions per day for 6 months.
  Arms: WorkStation Intervention Group
Behavioral: Usual Working Condition — Participants will be asked to continue working at their desk in their usual manner.
  Arms: Usual Working Condition Group

SUMMARY:
This is a pilot study to assess the feasibility of using treadmill desks (Workstations) within a Louisiana office workplace and to determine the effects of walking while working in overweight or obese, sedentary individuals.

DETAILED DESCRIPTION:
Eligible participants will be randomized by chance to the WorkStation Intervention Group or to a Usual Working Condition Group.

The WorkStation Intervention Group will be asked to walk for up to 1.5 hours per day during the work week of Monday through Friday on the treadmill. Participants will complete two sessions per day for up to 45 minutes per session, tracking time and speed.

Usual Working Condition Group will be asked to continue working in usual environment and accustomed manner.

Regardless of which group the participants are assigned to, the participants will be asked to complete baseline and follow up assessment visits. Months 3 and 6 for approximately 1 hour for Body measurements (height, weight and waist circumference), body fat percent, gait speed, questionnaires, and accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* BMI ≥ 25 kg/m2
* Willing to give informed consent
* Willing to accept randomization to group assignment and willing to follow the protocol for the group to which they have been assigned
* Willing to maintain fulltime employment at the company for the next 6 months
* Willing to receive frequent contacts and communication from study staff over the next 6 months

Exclusion Criteria:

* Current participation in other Pennington Biomedical research studies
* BMI < 25 kg/m2
* Type 1 diabetes
* Average step count of ≥ 7,500 steps/day
* Self-reporting exercising > 20 minutes on 3 or more days/wk, within the past 6 months
* Unable to walk 45 minutes continuously without taking a rest
* Unable to walk without the use of an assistive device, such as a cane or walker
* Have had a cardiovascular event (stroke or heart attack) in the past 6 months
* Have a pacemaker or any other internal electrical medical device
* Have been diagnosed with Schizophrenia or bipolar disorder
* Have any condition that would limit participation in a physical activity program
* Women who are pregnant, have been pregnant in the last 6 months, or are breastfeeding
* Actively participating in a weight loss program
* Plan to move out of the study area within the next 6 months or plan to be away from work for more than 4 weeks in the next 6 months
* Have another member of household participating in the study
* Have any condition, which, in the opinion of the investigator would impede competence or compliance or possibly hinder completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Waist | 6 months
  Waist circumference will decrease in workers assigned to the WorkStation working condition relative to the usual working condition.

SECONDARY OUTCOMES:
Weight Assessments | 6 months
  Weight will improve in workers assigned to the WorkStation Group relative to the Usual Working Condition Group.
Body Fat Percent | 6 months
  Body fat percent will improve in workers assigned to the WorkStation Group relative to the Usual Working Condition Group.
Accelerometry | 6 months
  Participants' activity level measured by the accelerometer will increase in workers assigned to the WorkStation Group relative to the Usual Working Condition Group.
Gait Speed | 6 months
  Participants' gait speed will improve in workers assigned to the WorkStation Group relative to the Usual Working Condition Group.
Stress | 6 months
  Participants' stress level will decrease in workers assigned to the WorkStation Group relative to the Usual Working Condition Group.
Fatigue | 6 months
  Participants' fatigue level will decrease in workers assigned to the WorkStation Group relative to the Usual Working Condition Group.
Quality of life Questionnaire | 6 months
  Participants' quality of life will improve in workers assigned to the WorkStation Group relative to the Usual Working Condition Group.

CONTACTS AND LOCATIONS:
Overall Officials: Catrine Tudor-Locke, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States